CLINICAL TRIAL: NCT02156583
Title: Frailty: Prevalence and Response to Left Ventricular Assist Device Therapy in Older Heart Failure Patients
Status: Completed | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Collaborators: Thoratec Corporation (Industry); National Skeletal Muscle Research Center (Unknown); Greater New York Geriatric Cardiology Consortium (Unknown)
Responsible Party: Sponsor
Other Study IDs: 14C.146
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Systolic Heart Failure
Keywords: Ventricular Assist Device; Skeletal Muscle; Frailty; Older adults
MeSH Terms: conditions — Heart Failure, Systolic; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older, left ventricular assist device: Older heart failure patients undergoing left ventricular assist device implantation

SUMMARY:
This is an observational study evaluating changes in frailty and associated impairments in older heart failure patients receiving left ventricular assist device therapy.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old or older
* Scheduled to undergo left ventricular assist device implantation at Thomas Jefferson University

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Unable to complete baseline frailty assessment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive heart failure patients 60 years old or older undergoing left ventricular assist device implantation.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in frailty following left ventricular assist device implantation | Baseline (prior to surgery); 10 days, 1 month, 3 months, and 6 months post-operatively
  Frailty will be assess based on the domains initially described by Fried and colleagues: weakness, low physical activity, unintentional weight loss, slowness and exhaustion. Additional frailty measures include the Short Physical Performance Battery (SPPB), as well as gait speed and hand grip strength as single item measures.

SECONDARY OUTCOMES:
Skeletal muscle size as measured by ultrasonography | Baseline (prior to surgery); 10 days and 3 months postoperatively

OTHER OUTCOMES:
Cognitive function measured by the Montreal Cognitive Assessment | Baseline; 3 and 6 months post-operatively

CONTACTS AND LOCATIONS:
Overall Officials: Gordon R Reeves, MD, MPT, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Maurer MS, Horn E, Reyentovich A, Dickson VV, Pinney S, Goldwater D, Goldstein NE, Jimenez O, Teruya S, Goldsmith J, Helmke S, Yuzefpolskaya M, Reeves GR. Can a Left Ventricular Assist Device in Individuals with Advanced Systolic Heart Failure Improve or Reverse Frailty? J Am Geriatr Soc. 2017 Nov;65(11):2383-2390. doi: 10.1111/jgs.15124. Epub 2017 Sep 21. PMID 28940248